Document: TDOC-0057803 Version: 1.0; CURRENT; Most-Recent; Effective

Status: Effective

#### **Short Title:**

## Statistical Analysis Plan CLE383-P004 / NCT04528017

#### **Full Title:**

# Statistical Analysis Plan CLE383-P004

**Protocol Title:** Clinical Comparison of 2 Daily Disposable Contact Lenses –

Pilot Study 2

Protocol TDOC Number: TDOC-0057749

Job Notes:

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

Effective Date: 14-Aug-2020 Alcon - Business Use Only Statistical Analysis Plan

Version: 1.0; CURRENT; Most-Recent; Effective **Document:** TDOC-0057803

Status: Effective

**Executive Summary:** 

Key Objective:

The primary objective of this study is to evaluate the overall performance of PRECISION1<sup>TM</sup> (verofilcon A) Soft Contact Lenses (PRECISION1) when compared to CooperVision® Clariti® 1 day (Clariti 1-Day).

Decision Criteria for Study Success:

Decision criteria for study success are not applicable for this study.

Print Date: Printed By:

 ${\bf Alcon \textbf{-} Business} \ Use \ Only \ {\tt Statistical} \ {\tt Analysis} \ {\tt Plan}$ 

Effective Date: 14-Aug-2020 Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0057803

Status: Effective

## **Table of Contents**

| Statistic | al Analysis Plan CLE383-P004 | 1 |
|-----------|-----------------------------------------------------|----|
| Table of | f Contents | 3 |
| List of 7 | Tables | 4 |
| 1 | Study Objectives and Design | 5 |
| 1.1 | Study Objectives | |
| 1.2 | Study Description | 5 |
| 1.3 | Randomization | |
| 1.4 | Masking | 6 |
| 2 | Analysis Sets | 6 |
| 2.1 | Safety Analysis Set | 6 |
| 3 | Subject Characteristics and Study Conduct Summaries | 7 |
| 4 | Effectiveness Analysis Strategy | 7 |
| 4.1 | Effectiveness Endpoints | 7 |
| 4.2 | Effectiveness Hypotheses | 8 |
| 4.3 | Statistical Methods for Effectiveness Analyses | 9 |
| 4.3.1 | Primary Effectiveness Analyses | 9 |
| 5 | Safety Analysis Strategy | Q |
| 5.1 | Safety Endpoints | |
| 5.2 | Safety Hypotheses | |
| 5.3 | Statistical Methods for Safety Analyses | |
| 5.3.1 | Adverse Events | |
| 5.3.2 | Biomicroscopy Findings | |
| 5.3.3 | Device Deficiencies | |
| 6 | Sample Size and Power Calculations | |
| 7 | References | 11 |

| Alcon - Bus | siness Use Only Statistical Analysis Plan | Effective Date: 14-Aug-2020 |
|---|---|---|
| | Version: 1.0; CURRENT; Most | -Recent; Effective |
| Status: Effec | tive | |
| 8 | Revision History | 11 |
| 9 | Appendix | 12 |
| | List of Tables | |
| Table 1–1 | Study Description Summary | 5 |
| Table 10–1 | Overview of Study Plan | 12 |


Status: Effective

# 1 Study Objectives and Design

# 1.1 Study Objectives

#### **PRIMARY OBJECTIVE**

The primary objective of this study is to evaluate the overall performance of PRECISION1 contact lenses when compared to Clariti 1-Day.

## 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1 Study Description Summary

| Study Design | Prospective, randomized, bilateral, parallel group, crossover, |
|---|---|
| | double-masked, |
| Study Population | Volunteer subjects aged 18 or over who are habitual |
| | spherical soft contact lens wearers (excluding |
| | current/previous PRECISION1, Clariti 1-Day and DAILIES |
| | TOTAL1® lens wearers), have at least 3 months of contact |
| | lens wearing experience, and who wear their habitual lenses |
| | at least 5 days per week and at least 10 hours per day. |
| | Target to complete: 52 |
| | Planned to enroll: ~72 |
| Number of Sites | ~4 |
| | US |
| Test Product | PRECISION1 (verofilcon A) Soft Contact Lenses |
| | (PRECISION1) |
| Control Product | CooperVision® Clariti® 1 day (Clariti 1-Day) |
| Duration of Treatment | ~ 16 days total duration (test and control) |
| | Test Product: ~ 8 days |
| | Control Product: ~ 8 days |


Status: Effective

| Visits | Visit 1 (Day 0) – Screening/Baseline/Dispense Lens 1 |
|--------|-------------------------------------------------------------|
| | Visit 2 [Day 8 (-0/+3 Days)] – Week 1 Follow-up Lens |
| | 1/Dispense Lens 2 |
| | Visit 3 [Day 8 (-0/+3 Days)] – Week 1 Follow-up Lens 2/Exit |

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens sequence assignment. Randomization will be implemented in the Electronic Data Capture (EDC)/randomization integration system.

### 1.4 Masking

The study is double-masked.

# 2 Analysis Sets

# 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study.

. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

Subjects who are lost to follow-up and their exposure to dispensed study lenses is unknown will be included in the safety analysis data set.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.


Status: Effective

## 3 Subject Characteristics and Study Conduct Summaries

The following tables will be presented:

- Subject Disposition by Lens Sequence
- Analysis Set by Lens
- Analysis Set by Lens Sequence
- Subject Accounting by Lens Sequence
- Demographics Characteristics by Lens Sequence
- Baseline Demographics Characteristics by Lens Sequence

In addition, the following subject listings will be provided:

- Listing of Subjects Excluded from Protocol Defined Analysis Set
- Listing of Lens Sequence Assignment by Investigator
- Listing of Subjects Discontinued from Study

### 4 Effectiveness Analysis Strategy

The Safety

Analysis Set will be used for all effectiveness analyses.

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized with counts and percentages from each category.

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out.

# 4.1 Effectiveness Endpoints

#### **Primary Endpoint**

The primary endpoint is distance visual acuity (VA) with study lenses, collected in logMAR, for each eye.

Version: 1.0; CURRENT; Most-Recent; Effective **Document:** TDOC-0057803 Status: Effective **Effectiveness Hypotheses** 4.2 **Primary Effectiveness** No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.

Alcon - Business Use Only Statistical Analysis Plan

Effective Date: 14-Aug-2020


Status: Effective

# 4.3 Statistical Methods for Effectiveness Analyses

## 4.3.1 Primary Effectiveness Analyses



# 5 Safety Analysis Strategy

The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters. Therefore, no inferential testing will be done for the safety analysis.

# **5.1** Safety Endpoints

The safety endpoints are

Adverse events (AE)

Biomicroscopy findings

- Limbal hyperemia
- o Bulbar hyperemia
- Corneal staining
- Conjunctival staining
- Palpebral conjunctival observations
- Corneal epithelial edema


Status: Effective

- o Corneal stromal edema
- Corneal vascularization
- Conjunctival compression/indention
- o Chemosis
- Corneal infiltrates
- o Other findings

Device deficiencies

## 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

## 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses, Visit 1 for Period 1 and Visit 2 for Period 2. Safety variables will be summarized descriptively.

#### 5.3.1 Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.



The following tables and supportive listings will be provided:

- Incidence of All Ocular Treatment-Emergent Adverse Events
- Incidence of All Nonocular Treatment-Emergent Adverse Events
- Listing of All Ocular Treatment-Emergent Adverse Events
- Listing of All Nonocular Treatment-Emergent Adverse Events
- Listing of All Ocular Pre-Treatment Adverse Events


Status: Effective

• Listing of All Nonocular Pre-Treatment Adverse Events



## 5.3.2 Biomicroscopy Findings

The following tables and supportive listings will be provided:

- Frequency and Percentage for Biomicroscopy Findings by Visit
- Incidence of Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listing of Subjects With Other Biomicroscopy Findings
- Listing of Subjects With Increased Severity by 1 Grade in Biomicroscopy Findings
- Listing of Subjects With Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listings of Subjects with Infiltrates

#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure

## **6** Sample Size and Power Calculations

No formal sample size calculation is provided given the descriptive and pilot nature of the study.

#### 7 References

Not Applicable.

# **8** Revision History

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

#### Appendix 9

Overview of Study Plan **Table 10–1** 

| Procedure / Assessment | | Visit 1<br>Screening/Baseline/<br>Dispense Lens 1 | Visit 2<br>Week 1 Follow-up<br>Lens 1 □ / Dispense<br>Lens 2 | Visit 3<br>Week 1 Follow-up<br>Lens 2 □ / Exit | Unscheduled<br>Visit / Early<br>Exit |
|---|---|---|---|---|---|
| | | Ħ | 8 -0/+3 days after Visit 1 | 8 -0/+3 days after Visit<br>2 | N/A |
| Informed Consent | - | <b>√</b> | - | - | - |
| Demographics | - | ✓ | - | - | - |
| Medical History | - | ✓ | ✓ | ✓ | ✓ |
| Concomitant Medications | - | <b>√</b> | ✓ | ✓ | ✓ |
| Inclusion/Exclusion | <u>-</u> | <u>√</u> | | | |
| | | | 1 | | |
| Riomicroscopy | | | | | |
| Biomicroscopy - | | <u>'</u> | | | <u> </u> |
| | Ī | | | <b>-</b> | |
| | ı | | I | I | |
| Randomize | - | ✓ | - | - | - |
| Dispense (provide) study lenses - | | ✓ | ✓ | - | (✔) |

Alcon - Business Use Only Statistical Analysis Plan Effective


Status: Effective

| VA (logMAR distance) with study lenses, | _ | _ | 1 | 1 | _ |
|---|---|---|---|---|---|
| OD, OS | _ | _ | • | • | _ |
| | | I | | | I |
| | | I | • | • | - |
| | I | | | | |
| | I | I | | | |
| | I | | | | I |
| AEs | - | ✓ | <b>✓</b> | ✓ | ✓ |
| Device Deficiencies | - | <b>√</b> | <b>✓</b> | <b>√</b> | <b>√</b> |
| Exit Form | - | (✓) | (✓) | (✓) | (✔) |

 $\square$  subjects will be required to wear the study lenses for 10 (-2/+6) hours at the follow-up visits;

Effective Date: 8/14/2020 12:06:58 PM

Alcon - Business Use Only Statistical Analysis Plan Document: TDOC-0057803 Version: 1.0; CURRENT; Status: Effective Version: 1.0; CURRENT; Most-Recent; Effective

Page 14


Status: Effective


Status: Effective


Status: Effective

# Signature Page for V-CLN-0005190 v1.0 $\,$



Signature Page for V-CLN-0005190 v1.0